CLINICAL TRIAL: NCT02071199
Title: Treatment of Human Gingivitis With Topical ACCS: a Two Week Safety Dose-ranging and Proof-of-principle Trial
Brief Title: Treatment of Human Gingivitis With Amnion-derived Cellular Cytokine Solution (ACCS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Noveome Biotherapeutics, formerly Stemnion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ST-04-13
Record Dates: First submitted 2014-02-21; First posted 2014-02-25 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Gingivitis
Keywords: Gingivitis; Periodontitis; ACCS
MeSH Terms: conditions — Gingivitis; Periodontitis | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low dose 0.3X ACCS (Experimental): 20 microliters of 0.3X ACCS per tooth is applied directly excluding third molars by dental professional daily Monday through Friday for two weeks
  Interventions: Drug: 0.3X ACCS
- High dose 1X ACCS (Experimental): 20 microliters of 1X ACCS per tooth is applied directly excluding third molars by dental professional daily Monday through Friday for two weeks
  Interventions: Drug: 1X ACCS (Amnion-derived Cellular Cytokine Solution)
- Normal saline (Placebo Comparator): 20 microliters of saline placebo per tooth is applied directly excluding third molars by dental professional daily Monday through Friday for two weeks
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: 1X ACCS (Amnion-derived Cellular Cytokine Solution) — 1X ACCS will be applied to the gingival margin daily 5 days per week for 2 weeks
  Other Names: ACCS
  Arms: High dose 1X ACCS
Drug: Normal saline — Saline will be applied to the gingival margin daily 5 days per week for 2 weeks
  Other Names: saline placebo
  Arms: Normal saline
Drug: 0.3X ACCS — 0.3X ACCS will be applied to the gingival margin daily 5 days per week for 2 weeks
  Other Names: Diluted ACCS
  Arms: Low dose 0.3X ACCS

SUMMARY:
The purpose of this study is to evaluate the safety of oral topical application of Amnion-derived Cellular Cytokine Solution (ACCS) in subjects with gingivitis

DETAILED DESCRIPTION:
This randomized blinded study will evaluate the use of ACCS in subjects with gingivitis. Two doses of ACCS will be used. It will be given topically intra-orally daily Monday through Friday for 2 weeks. In the first cohort, a low dose of ACCS or saline will be given by random chance. If there are no safety issues, cohort two will include a higher dose of ACCS randomized with saline. Pocket depth, plaque index, gingival index, and bleeding on probing will be assessed. To assess shifts in supragingival flora, a qualitative and quantitative microbial analysis will be performed for common oral bacteria. There will also be an analysis of inflammatory cytokines in crevicular fluid at the beginning and end of the study. Comparisons of adverse events and outcomes will be made between the subjects receiving low dose ACCS, high dose ACCS, and saline.

ELIGIBILITY:
Inclusion Criteria:

* good general health
* ages 18-70 years
* minimum of 20 natural teeth
* modified gingival index score of 2.0 or greater and >40 percent bleeding sites at initial presentation.

Exclusion Criteria:

* presence of orthodontic appliance
* soft or hard tissue tumor of the oral cavity
* carious lesion requiring immediate treatment
* participation in another clinical trial within 30 days
* pregnant or breast-feeding women
* women of child-bearing potential refusing to use an acceptable method of birth control
* antibiotic therapy within the last 30 days
* chronic use (> 3 times/week) of non-steroidal anti-inflammatory medications (NSAID). Any use of steroids. Low dose (<325 mg) aspirin is allowed.
* immune-compromised subjects
* subjects with liver or kidney dysfunction on blood tests as evidenced by a value equal to or greater than 2X the upper limit of normal.
* any medical history or any concomitant medication that might affect the assessment of the study treatment or periodontal tissues such as diabetes rheumatoid arthritis, Crohn's disease, use of nifedipine, phenytoin (Dilantin), anticoagulant medications (e.g. warfarin), ongoing cancer treatment either with radiation of chemotherapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2014-03; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse/serious adverse events | End of two weeks of treatment and at two weeks follow-up visit

SECONDARY OUTCOMES:
Probing pocket depth | Bseline and after two weeks of treatment
  Depth will be measured at six sites per tooth
Modified gingival index | Baseline and after two weeks of treatment
  Gingival index will be measured at six sites per tooth
Bleeding on probing | Baseline and after two weeks of treatment
  Bleeding will be measured at six sites per tooth
Plaque index | Baseline and after two weeks of treatment
  Only the gingival third of the tooth will be evaluated
Microbial analysis | Baseline and after two weeks of treatment
  6 teeth will be sampled
Cytokine analysis | Baseline and after two weeks of therapy
  Inflammatory cytokines will be sampled in crevicular fluid

CONTACTS AND LOCATIONS:
Overall Officials: David L Steed, MD, Study Director — Noveome Biotherapeutics, formerly Stemnion
Locations (1):
- Forsyth Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No